CLINICAL TRIAL: NCT06579222
Title: Comorbidity Management in Rheumatic Disease: Assessing a Potential Care Gap in Patients With Rheumatoid Arthritis.
Brief Title: Comorbidity Management in Rheumatic Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Rheumatology Association (CIORA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 125677
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis; Comorbidities and Coexisting Conditions
Keywords: rheumatoid arthritis; comorbidities
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Comorbidity Clinic (Experimental): The following investigations and treatments will be offered as associated with a comprehensive comorbidity clinic appointment with the primary care rheumatology family physician: Blood pressure, heart rate, height and weight measurement. Blood work (standard lipid panel, fasting plasma glucose or glycated hemoglobin (A1C), eGFR, and Lipoprotein a, Bone densitometry (if applicable to the patient/participant).
  Vaccinations will be offered if applicable to the patient/participant according to Health Canada guidelines (Vaccination with Pneu-P-23, Pneu-C-13, herpes zoster and COVID-19 vaccine).
  Interventions: Other: Primary Care Rheumatology Family Physician Consultation

INTERVENTIONS:
Other: Primary Care Rheumatology Family Physician Consultation — The participant will be booked with a primary care rheumatology family physician for rheumatoid arthritis comorbidity screening. They will complete weight, height, blood pressure measurement, assess for risk factors for dyslipidemia, type 2 diabetes, hypertension, bone mineral density loss and vaccine preventable infectious diseases.

SUMMARY:
Rheumatoid arthritis is a disease where the immune system attacks the body by mistake, causing inflammation of the joints and other body parts. People with rheumatoid arthritis are at higher risk of infections, heart problems, and bone issues compared to others. They regularly see rheumatologists, arthritis care physicians, to manage their disease. However, managing these other health problems alongside their main treatment is difficult for rheumatologists due to limited resources. This clinical study is being conducted to see if adding a family doctor to a team of rheumatologists can help. Rheumatologists will complete a case report form about the patient's health and send them to a special family physician clinic. This clinic will focus on improving vaccination against diseases, heart health, and bone strength. They will check if patients need special vaccines to protect them from infections. They will screen for heart disease using blood pressure measurements, and order blood work for high cholesterol and diabetes if needed. They will also review bone health and send people for tests to check their bone density if needed. A change in routines and medications may be recommended after their checkup. Rheumatologists will complete another case report about the patient's health 6 months after their family doctor appointment. The study will assess how these markers of health management improve after this family doctor joins the team. It hopes to prove that this new way of working in the community will give people with rheumatoid arthritis better protection against certain infections, heart problems and weak bones.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Waterloo Rheumatology Community Clinic
* Aged 18 to 80 years of age
* Diagnosis of rheumatoid arthritis
* Minimum of limited working proficiency in English
* No significant cognitive impairment that can inhibit their ability to engage in the study

Exclusion Criteria:

* Age less than 18 years or greater than 80 years
* Significant cognitive impairment that impedes ability to engage in the study
* Unwilling to participate in the study
* Patients currently pregnant will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Care Gap: Pneumococcal vaccination | 6 months
  the number of care gaps (percentage of individuals who require treatment according to established guidelines, but do not receive it) identified and addressed within 6 months of comorbidity clinic intervention, for pneumococcal vaccination.
Care Gap: Cardiovascular screening | 6 months
  the number of care gaps (percentage of individuals who require treatment according to established guidelines, but do not receive it) identified and addressed within 6 months of comorbidity clinic intervention, for cardiovascular screening (determined by meeting a combination of blood pressure, cholesterol and blood sugar measurement guidelines)
Care Gap: Osteoporosis screening | 6 months
  The number of care gaps (percentage of individuals who require treatment according to established guidelines, but do not receive it) for osteoporosis prevention and screening (determined by meeting guidelines for Vitamin D supplementation and bone densitometry completion)

SECONDARY OUTCOMES:
Care Gap: vaccine-preventable diseases (herpes zoster, influenza and COVID-19) | 6 months
  the number of care gaps (percentage of individuals who require treatment according to established guidelines, but do not receive it) identified and managed for remaining vaccine-preventable diseases (herpes zoster, influenza and COVID-19).
Care Gap: Comorbidity treatment with medication | 6 months
  (percentage of individuals who require treatment according to established guidelines, but do not receive it) identified and managed for the initiation of antihypertensive agents, cholesterol-lowering medications or medications for type 2 diabetes in study participants within the 6 months following the comprehensive comorbidity clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Schulz, Principal Investigator — Western University
Locations (1):
- Waterloo Rheumatology, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No